CLINICAL TRIAL: NCT00752934
Title: Does Oral Baclofen Improve Care and Comfort in Spastic Children in Nursing Homes?
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Principal Investigator, Dr. Hilla Ben-Pazi, PI, Shaare Zedek Medical Center
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 59/08
Record Dates: First submitted 2008-09-15; First posted 2008-09-16 (Estimated); Last update posted 2018-12-31 (Actual); Status verified 2018-12

CONDITIONS: Cerebral Palsy
Keywords: nursing homes; children; ages 1-18 years; spastic quadriplegia
MeSH Terms: conditions — Cerebral Palsy; Quadriplegia | interventions — Baclofen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- group a (Experimental): Baclofen followed by Placebo
  Interventions: Drug: oral baclofen + placebo
- group b (Experimental): Placebo followed by Baclofen
  Interventions: Drug: placebo + oral baclofen

INTERVENTIONS:
Drug: oral baclofen + placebo — Group A will be given 13 weeks of oral baclofen followed by a 2-week non-treatment (washout) period, and then 13 weeks of oral placebo.
  For participants who with weight under 15 Kg at the time of enrolment, the initial oral baclofen dose will be 2.5 mg daily, increasing weekly over a 7-week period to 10 mg three times a day, and will be continued at that dose for the following 5 weeks.
  For those participants who will be over 15 Kg at the time of enrollment, the starting oral baclofen dose will be 5 mg daily, increasing over a 9-week period to 20 mg three times a day, and will be continued for the next 3 weeks at that dose. At the end of each 12-week period, the drug (either baclofen or placebo) will be tapered over 6 days.
  Children's carers will given information on possible side effects, and asked to contact one of the researchers if any adverse events occur.
  Arms: group a
Drug: placebo + oral baclofen — Group B will receive 13 weeks of oral placebo followed by 2-week nontreatment, and then 13 weeks of oral baclofen
  Arms: group b

SUMMARY:
Baclofen is a drug that reduces the muscle stiffness. In disabled children that have very stiff muscles, the stiffness and secondary changes in the joints may cause discomfort and pain. In this study we will check if treatment with Baclofen reduces pain in disabled children with stiff muscles.

ELIGIBILITY:
Inclusion Criteria:

* Cerebral palsy nursing homes children ages 1-18 years spastic quadriplegia

Exclusion Criteria:

* active epilepsy severe truncal hypotonia

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2010-10; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
care and comport questionnaires | 28 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Saare Zedek Medical Center, Jerusalem, Israel